CLINICAL TRIAL: NCT01331031
Title: Association Between Parafunctional Habits and Signs and Symptoms Temporomandibular Disorder in Adolescents
Brief Title: Parafunctional Habits and Temporomandibular Disorder in Adolescents
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Lara Jansiski Motta, UniNove
Other Study IDs: 013/2008
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2010-10

CONDITIONS: Temporomandibular Disorder; Adolescent Behavior
Keywords: temporomandibular disorder; adolescents
MeSH Terms: conditions — Temporomandibular Joint Disorders; Adolescent Behavior

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adolescents: Adolescents between 10 and 20 years of age and enrolled in a municipal school system.

SUMMARY:
The disorders that affect the temporomandibular joint (TMJ) are responsible for the diverse symptoms. Objective: To evaluate whether or not the relationship between signs or symptoms of TMD and presence of harmful habits. The investigators evaluated 244 adolescents enrolled in public school . The investigators used the questionnaire for selection of orofacial pain and temporomandibular disorders, recommended by American Academy of Orofacial Pain to assess the presence or absence of signs and symptoms of TMD.

DETAILED DESCRIPTION:
For the assessment of signs and symptoms of TMD and parafunctional habits, 244 adolescents between 10 and 20 years of age and enrolled in a municipal school system were analyzed. The participants were submitted to the self-explanatory questionnaire for screening recommended by the American Academy of Orofacial Pain for the determination of orofacial pain and TMD. This questionnaire is made up of ten guided questions with yes or no responses to the most frequent signs and symptoms of orofacial pain and TMD. According to the Academy, three or more affirmative responses are an indication of TMD. Patient history and a detailed clinical exam were performed for the assessment of the presence or absence of parafunctional habits.

The frequency of signs and symptoms was analyzed and the data were described based on gender and age. The SPSS 12.0 program was used for the statistical analysis and the data were treated using the chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* age: 10 to 20 years old

Exclusion Criteria:

* no signing a term of informed consent

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 244 adolescents between 10 and 20 years of age and enrolled in a municipal school system.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, Ms, Principal Investigator — University of Nove de Julho
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil